CLINICAL TRIAL: NCT06843876
Title: The Evaluation of the Prototype Digital Vaccine Platform "TM-VAX" Among User in the Hospital for Tropical Diseases
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Thundon Ngamprasertchai, MD, Associate Professor, Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MUTM 2025-003-01
Record Dates: First submitted 2025-02-18; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Evaluate the Prototype Digital Vaccine Platform

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Subgroup: Healthcare Provider and Patients (Experimental)
  Interventions: Other: digital vaccine platform "TM VAX" application

INTERVENTIONS:
Other: digital vaccine platform "TM VAX" application — Physicians and healthcare providers and Patients will use the TM-VAX system for at least one week. Investigators will distribute the online questionnaire via Jotform through the LINE application at day 7, which will take around 10-15 minutes to complete. If participants have any questions or encounter any issues with the questionnaire, the research team will provide assistance and answer questions via the LINE application or in-person

SUMMARY:
RATIONALE:

Digital technology plays a key role in modern healthcare, impacting diagnosis, treatment, and health information management. Vaccination is a critical tool for disease prevention, reducing healthcare costs, and enhancing quality of life. Managing vaccine records accurately is essential due to varying vaccine schedules and dosage requirements. Traditionally, paper-based vaccine records have faced challenges like loss, illegibility, and incomplete information. Digital solutions offer a more reliable method for managing vaccination data efficiently. A vaccine mobile application is a digital tool designed to improve record immunization by using mobile technology. These apps offer features like reliable vaccine information, immunization record tracking, and reminders for vaccinations. They also facilitate communication between individuals, healthcare providers, and public health systems, aiming to boost vaccine uptake and reduce hesitancy. Examples include ReadyVax offer evidence-based vaccine information to healthcare providers and patients, ImmunizeCA for managing immunization records in Canada, and MomsTalkShots, deliver tailored educational content to increase vaccine uptake among specific populations, like pregnant women. Some apps, like HANDI, assist in public health data management, while application SafeVac and v-safe monitor post-vaccination safety. In Thailand, apps like StatelessVac and RamaCovid have supported immunization efforts and Coronavirus disease 2019 (COVID-19) vaccination. Thus, advancing mobile health technologies are valuable tools for improving healthcare delivery and enhancing immunization practices in the modern era.

OBJECTIVE: To evaluate the prototype digital vaccine platform "TM-VAX" user by Technology Acceptance Model (TAM)

METHODOLOGY:

This is a single-center, cross-sectional study conducted in the Hospital for Tropical Diseases, Mahidol University, Bangkok, Thailand, between February and May 2025. The study will recruit 200 participants, divided into two groups: 30 healthcare providers and 170 patients. Participants will be allowed to use the TM-VAX application for a one-week trial. Data will be collected through a single online questionnaire (Jotform), with the researcher distributing the questionnaire link via the LINE application (if applicable) or in-person at the end of study (day7). Data collection takes time around 10-15 minutes. The questionnaire consists of three main parts: demographic data, usage experience, and satisfaction. The sections on usage and satisfaction were developed based on previous literature and validated tools such as the mHealth App Usability Questionnaire (MAUQ) and the Usefulness, Satisfaction, and Ease of Use (USE) Questionnaire. The investigators adapted the usage and satisfaction sections from the MAUQ, including 20 questions organized into two parts. Part 1 comprises four categories: Ease of Use (6 items), System Information and Functionality (5 items), Communication (3 items), and Satisfaction (6 items), which addresses overall user satisfaction. Responses are scored on a 5-point Likert scale, with a high score (5 points) indicating very high usage or satisfaction, and the lowest score (1 point) indicating low usage or satisfaction. Part 2 includes open-ended questions to gather users' opinions about a problem and obstacles in using the application, as well as suggestions for improvement. Some participants will be randomly selected to in-depth interview (if participants are willing to do so).

ELIGIBILITY:
Inclusion Criteria:

Healthcare Provider:

* Aged 18 years or older
* Thai nationality
* Currently working at the Hospital for Tropical Diseases, regardless of work duration
* Have basic skills in using computers, mobile phones, and the internet
* Willing to participate in the study

Patients:

* Aged 18 years or older
* Thai nationality
* Have basic skills in using computers, mobile phones and the internet
* Willing to participate in the study

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
User satisfaction score with the digital vaccine platform "TM-VAX" as measured by the Technology Acceptance Model (TAM) Questionnaire | 1 week

IPD SHARING:
Plan to Share IPD: No